CLINICAL TRIAL: NCT01782781
Title: Local Infiltration Analgesia After Abdominal Hysterectomy
Acronym: LIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIA-AH-1
Record Dates: First submitted 2013-01-07; First posted 2013-02-04 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2014-10

CONDITIONS: Pain
Keywords: Analgesia; Local infiltration analgesia; Pain, relief; Pain, Postoperative; Ropivacaine; Ketorolac; Epinephrine; Adrenergic Agonists; Sympathomimetics; Therapeutic Uses; Anti-Inflammatory Agents, Non-Steroidal; Analgesics, Non-Narcotic; Analgesics; Opioids; Morphine; Pain; Postoperative Complications; Physiological Effects of Drugs; Anesthetics, Local; Anesthetics
MeSH Terms: conditions — Pain; Agnosia; Pain, Postoperative; Postoperative Complications | interventions — Ropivacaine; Epinephrine; Ketorolac Tromethamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group P (Placebo Comparator): Group P (Placebo) receives a local infiltration of saline in the operating field and ketorolac iv.
  In Group P the injectant consists of saline, total volume 156 mL. This is infiltrated by the surgeon into the soft tissue of the vagina, tubosacral and rotundum ligaments, in the abdominal fascia and subcutaneous at the end of surgery. Ketorolac 30 mg (1 mL) is also injected iv.
  Interventions: Drug: Placebo
- Group A (Active Comparator): Group A (Active) receives a local infiltration of ropivacaine, ketorolac and epinephrine in the operating field and saline iv.
  Drug: ropivacaine, ketorelac and epinephrine
  In Group A the injectant mixture consists of ropivacaine 300 mg mixed with 30 mg ketorolac and 0.5 mg epinephrine, total volume 156 mL. This mixture is infiltrated by the surgeon into the soft tissue of the vagina, tubosacral and rotundum ligaments, in the abdominal fascia and subcutaneous at the end of surgery. One mL saline is also injected iv.
  Interventions: Drug: ropivacaine, ketorelac and epinephrine

INTERVENTIONS:
Drug: ropivacaine, ketorelac and epinephrine — Active group
  Other Names: Narop, Toradol and adrenaline
  Arms: Group A
Drug: Placebo — Placebo group
  Other Names: Saline
  Arms: Group P

SUMMARY:
The aim of the study is to evaluate traditional analgesic therapy after abdominal hysterectomy with single infiltration of local anesthetics in the surgical area at the end of surgery.

DETAILED DESCRIPTION:
The study is a controlled, double blind, prospective, randomized and performed at Sahlgrenska University Hospital in Goteborg, Sweden. The injectant mixture consists of 300 mg ropivacaine mixed with 30 mg ketorolac and 0.5 mg epinephrine. Total volume of the solution is 156 ml. The normal saline injection is used in the control group in the same manner as in the LIA group. The parameters which would be evaluated are consumption of morphine, pain intensity and side effects.

The primary objective is to evaluate whether local infiltration analgesia (LIA) into the operating field will reduce morphine consumption during the first 24 postoperative hours in patients undergoing abdominal hysterectomy (AH).

Secondary end-points are pain intensity, incidence of nausea and vomiting, sedation intensity.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring abdominal hysterectomy

Exclusion Criteria:

* Body mass index > 35
* American Society of Anesthesiologists classification > 3
* Renal dysfunction
* Allergic to acetylsalicylic acid
* Unwilling to provide informed consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 0-24 hours postoperatively

SECONDARY OUTCOMES:
Pain intensity (NRS, Numeric Rating Score 0-10) | 0-24 hours postoperatively
Incidence of nausea and vomiting | 0-24 hours postoperatively
Sedation intensity (Ramsey scale) | 0-24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Egron Thorn, MD, PhD, Principal Investigator — Dept. of Anesthesia and Intensive Care, Sahlgrenska University Hospital, Goteborg, Sweden; Anil Gupta, MD, PhD, Study Chair — Dept. of Anesthesia and Intensive Care, Orebro University Hospital, Orebro, Sweden; Ove Carlsson, MD, Study Chair — Dept. of Anesthesia and Intensive Care, Sahlgrenska University Hospital, Goteborg, Sweden; Karin Olausson, MD, Study Chair — Dept. of Anesthesia and Intensive Care, Sahlgrenska University Hospital, Goteborg, Sweden; Olof Eckre, MD, PhD, Study Chair — Dept. of Anesthesia and Intensive Care, Sahlgrenska University Hospital, Goteborg, Sweden; Sven-Erik Ricksten, MD,PhD, Study Chair — Dept. of Anesthesia and Intensive Care, Sahlgrenska University Hospital, Goteborg, Sweden; Fatma Backman, MD, Study Chair — Dept. of Gynecological Surgery, Orebro University Hospital, Orebro, Sweden; Elisabeth Stadberg, MD, Study Chair — Dept. of Gynecological Surgery, Sahlgrenska University Hospital, Goteborg, Sweden
Locations (1):
- Dept. of Gynecological Surgery and Anesthesia and Intensive Care, Sahlgrenska University Hospital, Gothenburg, Sweden